CLINICAL TRIAL: NCT06392451
Title: A Multi-Site Clinical Evaluation of the LIAISON NES FLU A/B, RSV, & COVID-19 and LIAISON PLEX Respiratory (RSP) Flex Assays in Symptomatic Patients in Australia
Brief Title: LIAISON NES Influenza (FLU) A/B, Respiratory Syncytial Virus (RSV), & Coronavirus Disease 2019 (COVID-19) in Symptomatic Patients in Australia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DiaSorin Molecular LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DSM-PROT-005190
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Influenza A; Influenza Type B; Coronavirus Disease 2019; Respiratory Syncytial Virus (RSV); Adenovirus; Enterovirus; Para Influenza; Bordetella Parapertussis Infection; Bordetella Pertussis Infection, Respiratory; Chlamydia Pneumonia; Mycoplasma Pneumonia
MeSH Terms: conditions — COVID-19; Adenoviridae Infections; Enterovirus Infections; Paramyxoviridae Infections; Whooping Cough; Psittacosis; Pneumonia, Mycoplasma

STUDY DESIGN:
Masking Description: Participants are not provided investigational results and will only be provided with routine standard of care diagnostics results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Blinded, Prospective Arm (Other): Clinical specimens shall be collected prospectively from patients with signs or symptoms of respiratory tract infection. Nasal swab (NS) in Copan universal transport media (UTM) 3 milliliters for comparator testing should be collected by a healthcare professional. Where subjects are willing and able, up to 40% of NS for the investigational device will be self-collected under the guidance and supervision of a healthcare professional.
  Nasopharyngeal (NPS) specimens (optional) should only be collected by a healthcare professional. All specimens collected from children 13 years or younger should only be collected by a trained healthcare professional. Follow the Centers for Disease Control and Prevention guidelines for collecting NPS swabs, unless otherwise specified by the sponsor.
  Interventions: Diagnostic Test: LIAISON NES FLU A/B, RSV, & COVID-19; Diagnostic Test: LIAISON PLEX Respiratory Flex Assay

INTERVENTIONS:
Diagnostic Test: LIAISON NES FLU A/B, RSV, & COVID-19 — The LIAISON® NES FLU A/B, RSV & COVID-19 real-time (RT) PCR assay is a Point of Care (POC) system that enables the extraction, amplification, detection and differentiation of influenza A, Influenza B, respiratory syncytial virus (RSV) and SARS-CoV-2 viral RNA from dry nasal swabs (NS). The system consists of the LIAISON® NES FLU A/B, RSV & COVID-19 cartridge, the LIAISON® NES system (with LIAISON® NES Software), and associated accessories. In the LIAISON® NES FLU A/B, RSV & COVID-19 cartridge, extraction reagents and lyophilized fluorescent probes are used together with corresponding forward and reverse primers to extract and amplify influenza A, influenza B, RSV, SARS-CoV-2 and internal control RNA targets.
Diagnostic Test: LIAISON PLEX Respiratory Flex Assay — The LIAISON PLEX® (also known as VERIGENE® II) RSP Flex Assay is an automated test for the detection and identification of common viruses and bacteria, including severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) RNA, from upper respiratory specimens. The VERIGENE® II Respiratory Flex (RSP Flex) Assay is performed on the VERIGENE® II System. The VERIGENE® II System is an automated platform that performs sample preparation and is capable of polymerase chain reaction (PCR) for the detection of target-specific nucleic acids. The VERIGENE® II System is a fully automated, bench-top "sample-to-answer" device. The test reagents are supplied in a single, disposable test cartridge.
  Other Names: VERIGENE II

SUMMARY:
To establish the relative accuracy of the LIAISON® NES Flu A/B, RSV & COVID-19 assay for viral nucleic acid targets from professionally collected or patient self-collected dry nasal (NS) swabs and to establish the relative accuracy of the LIAISON PLEX® RSP Flex assay from NS and nasopharyngeal swabs (NPS) in applicable transport media from human patients exhibiting clinical signs and symptoms of a respiratory tract infection.

DETAILED DESCRIPTION:
This study is a clinical evaluation of two investigational devices on the same patient specimens:

* The LIAISON® NES FLU A/B, RSV & COVID-19 assay used for the detection and identification of influenza A, influenza B, RSV and SARS-CoV-2 on the LIAISON® NES system, developed by DiaSorin Molecular
* The LIAISON PLEX® RSP Flex assay used for the detection and identification of 19 common respiratory pathogens, including 14 viral and 5 bacterial targets on the LIAISON PLEX® system, developed by Luminex Corporation (a subsidiary of DiaSorin)

This study will utilize untrained operators to perform investigational device testing on the LIAISON NES platform, and as such instrument or assay-specific training will not be provided beforehand. Sites will receive the necessary protocols and instructions for use required to implement the study protocol. Testing on the LIAISON PLEX® platform will be performed by trained operators. Study staff will receive training on the device prior to the start of testing. The diagnostic accuracy of the LIAISON® NES FLU A/B, RSV & COVID-19 assay will be evaluated using dry NS specimens prospectively collected from patients who meet the study inclusion criteria. The diagnostic accuracy of the LIAISON PLEX® RSP Flex assay will be evaluated using NS and NPS specimens prospectively collected from patients who meet the study inclusion criteria and stored in the applicable transport media. Performance of the LIAISON® NES FLU A/B, RSV & COVID-19 and LIAISON PLEX® RSP Flex assays will be compared to one or more US FDA-cleared molecular assays, or as required by the local regulatory body.

Approximately 600-1000 prospective specimens will be tested using the LIAISON® NES FLU A/B, RSV & COVID-19 and LIAISON PLEX® RSP Flex assays, with a goal to obtain approximately 50 comparator method confirmed positives per target for influenza A and SARS CoV-2 and 30 comparator method confirmed positives per target for influenza B and RSV. The study is estimated to be conducted for approximately 3 months and should cover the length of the flu season, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Human patients with active signs and symptoms of respiratory tract infection at time of collection
* Specimens collected within 7 days of symptom onset for the initial collection
* Patient consents to participate in the study
* Availability of age, gender, race, ethnicity, collection dates, collection time, routine respiratory testing method, routine respiratory result, signs and symptoms (e.g., fever), date of symptom onset for each symptom, vaccination status (Flu and COVID-19, as applicable), pre-existing medical conditions (as applicable), medications (e.g., COVID-19 antivirals), etc. for each subject

Exclusion Criteria:

* Incorrect swab type
* Incorrect transport media
* Incorrect specimen handling (specimens not stored at recommended temperature)
* Samples collected >7 days from symptom onset
* Subject does not provide informed consent or subject withdraws informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-05-06 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | Samples will be tested on LIAISON NES within one hour of collection.
  Estimates of Sensitivity/PPA and Specificity/NPA will be calculated based on a two-by-two table (comparator method result vs. result from LIAISON® NES FLU A/B, RSV & COVID-19 assay or LIAISON PLEX® RSP Flex assay) for each target. In addition, 95% two-sided confidence intervals will be provided. A separate Sensitivity/PPA and Specificity/NPA for each target, to include those specimens excluded due to a discrepancy between the standard-of-care and molecular comparator result, will be presented in a separate 2 x 2 table.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Farhang, PhD, Principal Investigator — DiaSorin Molecular/Luminex Corporation
Locations (4):
- Australia (4):
  - Key Health - Bondi, Bondi Junction, New South Wales
  - Key Health - CBD South, Sydney, New South Wales
  - Key Health - Pagewood, Sydney, New South Wales
  - Maxwell Medical Group, Melbourne, Victoria